CLINICAL TRIAL: NCT07008131
Title: Impact on Major Urologic Complications With Prophylactic Use of Double J Catheter in Extravesical Ureteroneocystostomy in Renal Transplant Recipients
Brief Title: Impact of Double J Catheter in Major Urological Complications in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, MD, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-2018-1001-201
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Urinary Complications; Double J Stent
Keywords: Kidney Transplant; Urinary Complications; Double J stent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double J catheter colocation (Experimental): Double J catheter colocation in extravesical ureteroneocystostomy
  Interventions: Device: Double J stent
- No double J catheter colocation (Active Comparator): Extravesical ureteroneocystostomy with no double J catheter colocation
  Interventions: Procedure: No Double J stent

INTERVENTIONS:
Device: Double J stent — Extravesical ureteroneocystostomy with double J-catheter placement
  Arms: Double J catheter colocation
Procedure: No Double J stent — Extravesical ureteroneocystostomy with no Double J stent colocation
  Arms: No double J catheter colocation

SUMMARY:
Renal transplantation is the renal replacement therapy of choice in patients with end-stage chronic kidney disease. Major urological complications such as urinary leakage, ureteral stricture and urinary tract infections are usually observed in the first three months post-transplantation and lead to higher morbidity and mortality and lower graft function.

To evaluate the use of the double J catheter on major urological complications in extravesical ureteroneocystostomy in renal recipients.

Open clinical trial. Renal transplant recipients were included, who underwent extravesical ureteroneocystostomy with trans-surgical placement of double J catheter compared to extravesical ureteroneocystostomy without trans-surgical catheter placement. The study variables were urinary leakage, ureteral stricture, urinary tract infection, surgical complications and graft function.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Renal transplantation candidates
* They agree to participate in the study

Exclusion Criteria:

* Previous renal transplantation
* Urinary tract malformations
* Urinary reservoir carriers
* Known neurogenic disease of the urinary tract
* Cadaveric donor grafts
* Grafts with double collecting system
* Patients whose trans-surgical findings require catheter placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Major urological complications | From enrollment to three months
  Urinary leakage, uretheral stenosis and urinary infection

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Biomédica 02, Hospital de Especialidades, Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No